CLINICAL TRIAL: NCT05411926
Title: Effect of PD-1 /PD-L1 Inhibitor Therapy Before Liver Transplantation on Acute Rejection After Liver Transplantation in Patients With Hepatocellular Carcinoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Tsinghua Chang Gung Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 21299-4-03
Record Dates: First submitted 2022-04-20; First posted 2022-06-09 (Actual); Last update posted 2022-06-09 (Actual); Status verified 2022-03

CONDITIONS: Hepatocellular Carcinoma; Acute Rejection
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — peripheral blood ， donor liver tissue， diseased liver tissue
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- The group that receiving PD-1 / PD-L1 inhibitor before liver transplantation
- The group without receiving PD-1 / PD-L1 inhibitor before liver transplantation

SUMMARY:
This study is a single-center, prospective, non-interventional cohort study based on the real world data.In this study, 30 patients with a history of PD-1/PD-L1 monotherapy prior to liver transplantation and 30 patients without a history of PD-1/PD-L1 monotherapy prior to liver transplantation were recruited from the group of patients with hepatocellular carcinoma who had undergone allogeneic liver transplantation.Collected patient data included demographics, oncology and immunotherapy history, evaluated index before liver transplantation, laboratory, pathological and imaging results at specific time points after transplantation (1 week, 2 weeks, 3 weeks, 4 weeks, 12 weeks, 16 weeks, 24 weeks), as well as the occurrence of acute rejection (AR) , grading of severity, and anti-rejection treatment plan at the same time. Endpoints included relapse-free survival and overall survival (OS). These data aims to assess: 1) the incidence of acute rejection after liver transplantation in patients with hepatocellular carcinoma; 2) the time of acute rejection, Banff classification, and acute rejection-related mortality after liver transplantation in patients with hepatocellular carcinoma; 3) the cellular immune function after liver transplantation;; 4) the dose and drug concentration of tacrolimus after liver transplantation in patients with hepatocellular carcinoma; and 5) the overall survival (OS) and relapse-free survival(RFS) after liver transplantation in patients with hepatocellular carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. age between 18 and 70 years,
2. Eastern Cooperative Oncology Group (ECOG) performance score ≤3,
3. voluntarily participate, totally understand in the study and sign the Informed Consent Form (ICF),
4. hepatopathology confirmed hepatocellular carcinoma after liver transplantation, 5）patients with hepatocellular carcinoma treated with PD1/PD-L1 monoclonal antibody prior to liver transplantation,

6）PD-1/PD-L1 monotherapy needs to be used ≥ 2 times (The patients were divided into observation and control group according to whether received PD-1/PD-L1 monoclonal antibody treatment before liver transplantation)

Exclusion Criteria:

1. patients with incomplete clinicopathological data,
2. post-transplantation ≥6months,
3. PD-1/PD-L1 monotherapy required for oncological reasons after liver transplantation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with hepatocellular carcinoma who had undergone allogeneic liver transplantation.In this study, 30 patients with a history of PD-1/PD-L1 monotherapy prior to liver transplantation and 30 patients without a history of PD-1/PD-L1 monotherapy prior to liver transplantation were recruited from the group of patients with hepatocellular carcinoma who had undergone allogeneic liver transplantation.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-03-17 (Actual); Primary Completion 2023-03 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
1) the incidence of acute rejection after liver transplantation in patients with hepatocellular carcinoma; | 2021-03~2023-03
2) the severity of acute rejection after liver transplantation in patients with hepatocellular carcinoma; | 2021-03~2023-03
3) the cellular immune function after liver transplantation，including lymphocyte subsets and cytokines | 2021-03~2023-03
4) the dose and drug concentration of tacrolimus after liver transplantation in patients with hepatocellular carcinoma; | 2021-03~2023-03

SECONDARY OUTCOMES:
5) the overall survival (OS) and relapse-free survival(RFS) after liver transplantation in patients with hepatocellular carcinoma. | 2021-03~2023-03

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tsinghua Changgung Hospital, Beijing, Beijing Municipality, China